CLINICAL TRIAL: NCT00723073
Title: Evaluation of Caspofungin or Micafungin as Empiric Antifungal Therapy in Adult Patients With Persistent Febrile Neutropenia: A Retrospective, Observational, Sequential Cohort Analysis
Brief Title: Caspofungin or Micafungin as Empiric Antifungal Therapy for Persistent Fever and Neutropenia
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: David W, Kubiak, PharmD, BCPS / Infectious Disease Clinical Specialist, Brigham and Women's Hospital
Other Study IDs: 2008-P-000605/1; BWH
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Results first posted 2010-08-04 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Febrile Neutropenia
Keywords: micafungin, caspofungin, febrile neutropenia
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Caspofungin arm: All patients admitted to BWH/DFCI who received at least 2 doses of caspofungin with an Absolute Neutrophil Count (ANC) < 500, for persistent febrile neutropenia from 11/1/2005 - 10/31/2006, as there first antifungal agent.
- Micafungin arm: All patients admitted to BWH/DFCI who received at least 2 doses of micafungin with an Absolute Neutrophil Count (ANC) < 500 for persistent febrile neutropenia from 11/1/2006 - 10/31/2007 as there first antifungal agent

SUMMARY:
Invasive fungal infections are an important cause of morbidity and mortality in patients with neutropenia who are receiving chemotherapy for cancer. Early diagnosis of these infections is difficult and fever may be the only sign. A delay in treatment while a diagnosis is pursued may lead to increased morbidity and mortality. There are now several echinocandins available with similar in vitro spectrum of activity. Caspofungin is the only echinocandin Food and Drug Administration (FDA) approved for empiric antifungal therapy in febrile neutropenia. Although all echinocandin antifungal agents have similar spectrum of activity, there are limited data on the use of micafungin in patients with persistent fever and neutropenia (FN). In November 2006 the Pharmacy and Therapeutics Committee at Brigham & Women's Hospital / Dana Farber Cancer Institute (BWH/DFCI) switched from caspofungin to micafungin as our formulary echinocandin. Given the limited clinical data on the use of micafungin as empiric antifungal therapy in patients with FN, we sought to evaluate the safety and effectiveness of micafungin, compared with caspofungin, for this indication using a sequential cohort analysis of patients treated before and after the formulary change at Brigham and Women's Hospital.

DETAILED DESCRIPTION:
Objectives

This retrospective cohort analysis of converting from caspofungin to micafungin as empiric antifungal therapy for cancer patients who are persistently febrile and neutropenic after receiving broad spectrum antibiotics at Brigham & Women's Hospital / Dana Farber Cancer Institute (BWH/DFCI) is designed to evaluate the following objectives:

* Safety of micafungin in this patient population
* Effective dose of 100 mg daily of micafungin compared to 70mg x1, then 50 mg daily of caspofungin
* Economic impact of converting or formulary echinocandin from micafungin to caspofungin

Study Design

* Retrospective cohort analysis - limited to medical records
* Data to be collected include the following:

  * Demographic information: including: gender, age, race
  * Past medical history and admitting diagnoses
  * Laboratory results: Liver function tests (LFTs), Including alanine aminotransferase (ALT), aspartate aminotransferase (AST), Total bilirubin, as well as serum fungal assays: Serum Galactomannan assay, 1.3-BD Glucan assay
  * Concomitant medications and duration of therapy for all systemic: antibiotics and antifungals
  * All invasive breakthrough fungal infection details, including speciation and outcomes during echinocandin therapy
  * Dosing, duration, and adverse events associated with echinocandin therapy

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to BWH/DFCI who received at least 2 doses of caspofungin with an Absolute Neutrophil Count (ANC) < 500, for persistent febrile neutropenia from 11/1/2005 - 10/31/2006, as there first antifungal agent.
* All patients admitted to BWH/DFCI who received at least 2 doses of micafungin with an Absolute Neutrophil Count (ANC) < 500 for persistent febrile neutropenia from 11/1/2006 - 10/31/2007 as there first antifungal agent

Exclusion Criteria:

* Patients receiving an echinocandin antifungal agent (micafungin or caspofungin) for an indication other then empiric therapy in febrile neutropenia
* Patients receiving therapy for an active or on-going invasive fungal infection
* Patients who received both caspofungin and micafungin during the same admission
* Patients with an ANC > 500 at when either micafungin or caspofungin was started
* Patients who received another antifungal agent for persistent febrile neutropenia, e.g., voriconazole, amphotericin B liposome, posaconazole, etc... Before they received an echinocandin (caspofungin or micafungin) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients who are persistently febrile and neutropenic after receiving broad spectrum antibiotics and receive empiric antifungal therapy with either caspofungin or micafungin
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Kubiak, PharmD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Schuler U, Bammer S, Aulitzky WE, Binder C, Bohme A, Egerer G, Sandherr M, Schwerdtfeger R, Silling G, Wandt H, Glasmacher A, Ehninger G. Safety and efficacy of itraconazole compared to amphotericin B as empirical antifungal therapy for neutropenic fever in patients with haematological malignancy. Onkologie. 2007 Apr;30(4):185-91. doi: 10.1159/000100055. Epub 2007 Mar 23. PMID 17396041
- [Background] Toubai T, Tanaka J, Ota S, Shigematsu A, Shono Y, Ibata M, Hashino S, Kondo T, Kakinoki Y, Masauzi N, Kasai M, Iwasaki H, Kurosawa M, Asaka M, Imamura M. Efficacy and safety of micafungin in febrile neutropenic patients treated for hematological malignancies. Intern Med. 2007;46(1):3-9. doi: 10.2169/internalmedicine.46.6021. Epub 2007 Jan 1. PMID 17202726
- [Background] Seibel NL, Schwartz C, Arrieta A, Flynn P, Shad A, Albano E, Keirns J, Lau WM, Facklam DP, Buell DN, Walsh TJ. Safety, tolerability, and pharmacokinetics of Micafungin (FK463) in febrile neutropenic pediatric patients. Antimicrob Agents Chemother. 2005 Aug;49(8):3317-24. doi: 10.1128/AAC.49.8.3317-3324.2005. PMID 16048942
- [Background] Walsh TJ, Teppler H, Donowitz GR, Maertens JA, Baden LR, Dmoszynska A, Cornely OA, Bourque MR, Lupinacci RJ, Sable CA, dePauw BE. Caspofungin versus liposomal amphotericin B for empirical antifungal therapy in patients with persistent fever and neutropenia. N Engl J Med. 2004 Sep 30;351(14):1391-402. doi: 10.1056/NEJMoa040446. PMID 15459300
- [Background] Walsh TJ, Pappas P, Winston DJ, Lazarus HM, Petersen F, Raffalli J, Yanovich S, Stiff P, Greenberg R, Donowitz G, Schuster M, Reboli A, Wingard J, Arndt C, Reinhardt J, Hadley S, Finberg R, Laverdiere M, Perfect J, Garber G, Fioritoni G, Anaissie E, Lee J; National Institute of Allergy and Infectious Diseases Mycoses Study Group. Voriconazole compared with liposomal amphotericin B for empirical antifungal therapy in patients with neutropenia and persistent fever. N Engl J Med. 2002 Jan 24;346(4):225-34. doi: 10.1056/NEJM200201243460403. PMID 11807146
- [Background] Wingard JR, White MH, Anaissie E, Raffalli J, Goodman J, Arrieta A; L Amph/ABLC Collaborative Study Group. A randomized, double-blind comparative trial evaluating the safety of liposomal amphotericin B versus amphotericin B lipid complex in the empirical treatment of febrile neutropenia. L Amph/ABLC Collaborative Study Group. Clin Infect Dis. 2000 Nov;31(5):1155-63. doi: 10.1086/317451. Epub 2000 Nov 7. PMID 11073745
- [Background] Winston DJ, Hathorn JW, Schuster MG, Schiller GJ, Territo MC. A multicenter, randomized trial of fluconazole versus amphotericin B for empiric antifungal therapy of febrile neutropenic patients with cancer. Am J Med. 2000 Mar;108(4):282-9. doi: 10.1016/s0002-9343(99)00457-x. PMID 11014720
- [Background] Walsh TJ, Finberg RW, Arndt C, Hiemenz J, Schwartz C, Bodensteiner D, Pappas P, Seibel N, Greenberg RN, Dummer S, Schuster M, Holcenberg JS. Liposomal amphotericin B for empirical therapy in patients with persistent fever and neutropenia. National Institute of Allergy and Infectious Diseases Mycoses Study Group. N Engl J Med. 1999 Mar 11;340(10):764-71. doi: 10.1056/NEJM199903113401004. PMID 10072411
- [Background] Ascioglu S, Rex JH, de Pauw B, Bennett JE, Bille J, Crokaert F, Denning DW, Donnelly JP, Edwards JE, Erjavec Z, Fiere D, Lortholary O, Maertens J, Meis JF, Patterson TF, Ritter J, Selleslag D, Shah PM, Stevens DA, Walsh TJ; Invasive Fungal Infections Cooperative Group of the European Organization for Research and Treatment of Cancer; Mycoses Study Group of the National Institute of Allergy and Infectious Diseases. Defining opportunistic invasive fungal infections in immunocompromised patients with cancer and hematopoietic stem cell transplants: an international consensus. Clin Infect Dis. 2002 Jan 1;34(1):7-14. doi: 10.1086/323335. Epub 2001 Nov 26. PMID 11731939
- [Background] Hughes WT, Armstrong D, Bodey GP, Bow EJ, Brown AE, Calandra T, Feld R, Pizzo PA, Rolston KV, Shenep JL, Young LS. 2002 guidelines for the use of antimicrobial agents in neutropenic patients with cancer. Clin Infect Dis. 2002 Mar 15;34(6):730-51. doi: 10.1086/339215. Epub 2002 Feb 13. No abstract available. PMID 11850858
- [Background] Vartivarian SE, Anaissie EJ, Bodey GP. Emerging fungal pathogens in immunocompromised patients: classification, diagnosis, and management. Clin Infect Dis. 1993 Nov;17 Suppl 2:S487-91. doi: 10.1093/clinids/17.supplement_2.s487. PMID 8274615
- [Background] Perfect JR, Dodds Ashley E, Drew R. Design of aerosolized amphotericin b formulations for prophylaxis trials among lung transplant recipients. Clin Infect Dis. 2004 Oct 15;39 Suppl 4:S207-10. doi: 10.1086/421958. PMID 15546119
- [Background] Pfaller MA, Boyken L, Hollis RJ, Kroeger J, Messer SA, Tendolkar S, Diekema DJ. In vitro susceptibility of invasive isolates of Candida spp. to anidulafungin, caspofungin, and micafungin: six years of global surveillance. J Clin Microbiol. 2008 Jan;46(1):150-6. doi: 10.1128/JCM.01901-07. Epub 2007 Nov 21. PMID 18032613
- [Background] Kuse ER, Chetchotisakd P, da Cunha CA, Ruhnke M, Barrios C, Raghunadharao D, Sekhon JS, Freire A, Ramasubramanian V, Demeyer I, Nucci M, Leelarasamee A, Jacobs F, Decruyenaere J, Pittet D, Ullmann AJ, Ostrosky-Zeichner L, Lortholary O, Koblinger S, Diekmann-Berndt H, Cornely OA; Micafungin Invasive Candidiasis Working Group. Micafungin versus liposomal amphotericin B for candidaemia and invasive candidosis: a phase III randomised double-blind trial. Lancet. 2007 May 5;369(9572):1519-1527. doi: 10.1016/S0140-6736(07)60605-9. PMID 17482982
- [Background] Yanada M, Kiyoi H, Murata M, Suzuki M, Iwai M, Yokozawa T, Baba H, Emi N, Naoe T. Micafungin, a novel antifungal agent, as empirical therapy in acute leukemia patients with febrile neutropenia. Intern Med. 2006;45(5):259-64. doi: 10.2169/internalmedicine.45.1498. Epub 2006 Apr 3. PMID 16595990
- [Background] Pappas PG, Rotstein CM, Betts RF, Nucci M, Talwar D, De Waele JJ, Vazquez JA, Dupont BF, Horn DL, Ostrosky-Zeichner L, Reboli AC, Suh B, Digumarti R, Wu C, Kovanda LL, Arnold LJ, Buell DN. Micafungin versus caspofungin for treatment of candidemia and other forms of invasive candidiasis. Clin Infect Dis. 2007 Oct 1;45(7):883-93. doi: 10.1086/520980. Epub 2007 Aug 29. PMID 17806055
- [Background] Sucher AJ, Chahine EB, Balcer HE. Echinocandins: the newest class of antifungals. Ann Pharmacother. 2009 Oct;43(10):1647-57. doi: 10.1345/aph.1M237. Epub 2009 Sep 1. PMID 19724014
- [Result] Kubiak DW, Bryar JM, McDonnell AM, Delgado-Flores JO, Mui E, Baden LR, Marty FM. Evaluation of caspofungin or micafungin as empiric antifungal therapy in adult patients with persistent febrile neutropenia: a retrospective, observational, sequential cohort analysis. Clin Ther. 2010 Apr;32(4):637-48. doi: 10.1016/j.clinthera.2010.04.005. PMID 20435233

RESULTS

PARTICIPANT FLOW:
Groups:
- Caspofungin Arm: All patients admitted to BWH/DFCI who received at least 2 doses of caspofungin with an ANC < 500, for persistent febrile neutropenia from 11/1/2005 - 10/31/2006, as there first antifungal agent.
- Micafungin Arm: All patients admitted to BWH/DFCI who received at least 2 doses of micafungin with an ANC < 500 for persistent febrile neutropenia from 11/1/2006 - 10/31/2007 as there first antifungal agent
Period: Overall Study
Arm/Group | Caspofungin Arm | Micafungin Arm
Started | 149 | 174
Completed | 149 | 174
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caspofungin Arm | Micafungin Arm | Total
Number analyzed (Participants) | 149 | 174 | 323
Age Continuous [Median (Inter-Quartile Range); unit: years] | 49 [39 to 58] | 49 [40 to 58] | 49 [39 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 75 | 144
  Male | 80 | 99 | 179
Primary Underlying Disease [Number; unit: participants] — primary oncological diagnosis
  participants
    Acute myelogenous leukemia | 76 | 82 | 158
    Non-Hodgkin's lymphoma | 28 | 25 | 53
    Acute lymphoblastic leukemia | 9 | 20 | 29
    Hodgkin's lymphoma | 8 | 12 | 20
    Chronic myelogenous leukemia | 6 | 8 | 14
    Multiple myeloma | 6 | 8 | 14
    Myelodysplastic syndrome | 5 | 7 | 12
    Aplastic anemia | 3 | 5 | 8
    other onocological diagnosis | 8 | 7 | 15
hematopoietic stem cell transplantation status [Number; unit: participants]
  Hematopoietic stem cell transplantation | 81 | 108 | 189
  No - Hematopoietic stem cell transplantation | 68 | 66 | 134
Patient Weight, kg [Median (Inter-Quartile Range); unit: kilograms] | 80 [67 to 89] | 80 [65 to 95] | 80 [65 to 95]

OUTCOME MEASURES:

1. Primary Outcome: Composite Primary Endpoint: Number of Participants With an Overall Favorable Response to Echinocandin Therapy for Empiric Antifungal Therapy for Persistent Febrile Neutropenia (FN)
Description: Overall favorable response was defined as achievement of successful treatment of baseline fungal infections, survival to hospital discharge, absence of breakthrough Ivasive fungal disese (IFD), and lack of advserse events (AE) attributable to treatment that led to discontinuation of echinocandin therapy.
Time Frame: 11/1/2005 - 10/31/2007
Measure: Number; unit: participants
Arm/Group | Caspofungin Arm | Micafungin Arm
Number analyzed (Participants) | 149 | 174
participants
  Yes | 122 | 141
  No | 27 | 33
Statistical Analysis 1: Comparison: Caspofungin Arm vs Micafungin Arm; Test type: Superiority or Other; p = 0.96, Fisher Exact; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.89 to 1.10], Standard Deviation 1

2. Primary Outcome: Successful Treatment of Any Baseline Invasive Fungal Disease (IFD)
Description: Possible or proven baseline invasive fungal disease were defined as were diagnosed within the 2 days of initiating echinocandin therapy for persistent febrile neutropenia
Time Frame: 11/1/2005 - 10/31/2007
Measure: Number; unit: participants
Arm/Group | Caspofungin Arm | Micafungin Arm
Number analyzed (Participants) | 149 | 174
participants
  No Baseline IFD | 146 | 168
  Successfully treated baseline IFD | 2 | 4
  Unsuccessfully treated baseline IFD | 1 | 2
Statistical Analysis 1: Comparison: Caspofungin Arm vs Micafungin Arm; Test type: Superiority or Other; p > 0.99, Fisher Exact; Risk Ratio (RR) = 1.0, 95% CI 2-sided [0.38 to 2.70], Standard Deviation 1

3. Primary Outcome: Mortality at Hospital Discharge
Description: We assessed all patients in the study cohort who dischaged from the hospital alive
Time Frame: 11/1/2005 - 10/31/2007
Measure: Number; unit: participants
Arm/Group | Caspofungin Arm | Micafungin Arm
Number analyzed (Participants) | 149 | 174
participants
  Alive at hospital discharge | 137 | 161
  Died before hospitial discharge | 12 | 13
Statistical Analysis 1: Comparison: Caspofungin Arm vs Micafungin Arm; Test type: Superiority or Other; p > 0.99, Fisher Exact; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.44 to 1.97], Standard Deviation 1

4. Primary Outcome: Absence of Any Breakthrough Invasive Fungal Disease (IFD)
Description: a breakthrough invasive fungal disesase was defined as any fungal infection that was diagnosed > 3 days on or during therapy or within 7 days after completion of therapy with an echinocandin
Time Frame: 11/1/2005 - 10/31/2007
Measure: Number; unit: participants
Arm/Group | Caspofungin Arm | Micafungin Arm
Number analyzed (Participants) | 149 | 174
participants
  No breakthrough IFD | 133 | 153
  Breakthrough IFD | 16 | 21
Statistical Analysis 1: Comparison: Caspofungin Arm vs Micafungin Arm; Test type: Superiority or Other; p = 0.48, Fisher Exact; Risk Ratio (RR) = 1.12, 95% CI 2-sided [0.61 to 2.07], Standard Deviation 1

5. Primary Outcome: Lack of an Adverse Drug Event (ADE) Attributable to Echinocandin (EC) Therapy That Led to Discontinuation of Therapy
Description: Defined as any advsere event directly attributable to echinocandin treatment that led to discontinuation of therapy or switch to alternative therapy
Time Frame: 11/1/2005 - 10/31/2007
Measure: Number; unit: participants
Arm/Group | Caspofungin Arm | Micafungin Arm
Number analyzed (Participants) | 149 | 174
participants
  No ADE | 146 | 172
  ADE which caused EC therapy discontinuation | 3 | 2
Statistical Analysis 1: Comparison: Caspofungin Arm vs Micafungin Arm; Test type: Superiority or Other; p = 0.57, Fisher Exact; Risk Ratio (RR) = 0.57, 95% CI 2-sided [0.10 to 3.37], Standard Deviation 1

6. Secondary Outcome: Duration of Echinocadin Therapy for Persistent Febrile Neutropenia (FN)
Description: median duration of therapy with an echinocandin (caspofungin or micafungin) for persistent febrile neutropenia (FN)
Time Frame: 11/1/2005 - 10/31/2007
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caspofungin Arm | Micafungin Arm
Number analyzed (Participants) | 149 | 174
days | 10 [6 to 18] | 9 [6 to 16]
Statistical Analysis 1: Comparison: Caspofungin Arm vs Micafungin Arm; Test type: Superiority or Other; p = 0.66, Chi-squared

7. Secondary Outcome: Liver Function Tests (LFTs) Elevated During or After Echinocandin Therapy
Description: aspartate aminotransferase (AST) or alanine aminotransferase (ALT)> 5x the upper limit of normal (ULN) or total bilirubin > 3x the upper limit of normal (ULN)
Time Frame: 11/1/2005 - 10/31/2007
Measure: Number; unit: participants
Arm/Group | Caspofungin Arm | Micafungin Arm
Number analyzed (Participants) | 149 | 174
participants
  No LFT elevations | 110 | 132
  AST > 5x upper limit of normal | 14 | 15
  ALT > 5x upper limit of normal | 10 | 9
  Total Bilirubin >3x upper limit of normal | 15 | 18

8. Secondary Outcome: Specific Type of Adverse Event That Resulted in Echinocandin (EC) Therapy Discontinuation
Description: The description of the adverse event that resulted in discontinuation of echinocandin (EC) therapy
Time Frame: 11/1/2005 - 10/31/2007
Measure: Number; unit: participants
Arm/Group | Caspofungin Arm | Micafungin Arm
Number analyzed (Participants) | 149 | 174
participants
  No Adverse Event requiring EC discontinuation | 146 | 172
  Rash | 2 | 1
  Liver function Test (LFT) increase | 0 | 1
  Anaphylaxis | 1 | 0

9. Secondary Outcome: Duration of Hospitization
Description: Median number of days patients were hospitalized during the study period
Time Frame: 11/1/2005 - 10/31/2007
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caspofungin Arm | Micafungin Arm
Number analyzed (Participants) | 149 | 174
days | 29 [24 to 38] | 28 [23 to 38]
Statistical Analysis 1: Comparison: Caspofungin Arm vs Micafungin Arm; Test type: Superiority or Other; p = 0.22, Fisher Exact

10. Secondary Outcome: Duration of Neutropenia
Description: Median number of days patients were neutropenic during the study period
Time Frame: 11/1/2005 - 10/31/2007
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caspofungin Arm | Micafungin Arm
Number analyzed (Participants) | 149 | 174
days | 20 [13 to 30] | 17 [13 to 28]
Statistical Analysis 1: Comparison: Caspofungin Arm vs Micafungin Arm; Test type: Superiority or Other; p = 0.11, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Caspofungin Arm | Micafungin Arm
Serious Adverse Events (participants affected / at risk) | 3/149 | 2/174
Other Adverse Events (participants affected / at risk) | 15/149 | 18/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caspofungin Arm (N=149) | Micafungin Arm (N=174)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Liver function test elevation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caspofungin Arm (N=149) | Micafungin Arm (N=174)
AST > 5x ULN (Hepatobiliary disorders) | 14 (14) | 15 (15)
ALT > 5x ULN (Hepatobiliary disorders) | 10 (10) | 9 (9)
Total Bilirubin > 3x ULN (Hepatobiliary disorders) | 10 (15) | 18 (18)

LIMITATIONS AND CAVEATS:
Retrospective, observational, sequential cohort study conducted at a single center. Only adult patients were treated at our institution, so these results cannot be extrapolated to a pediatric population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No